CLINICAL TRIAL: NCT04114812
Title: Student-centred Learning With Near-peer Tutoring Compared With a Standard Faculty-led Course for Undergraduate Training in Abdominal Ultrasound. A Multicentre Open-label Randomized Controlled Trial.
Brief Title: Near-peer Tutoring Compared With a Standard Faculty-led Course for Undergraduate Training in Abdominal Ultrasound.
Acronym: SIGNATURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UBern SIGNATURE
Record Dates: First submitted 2019-09-27; First posted 2019-10-03 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Ultrasonography; Educational Techniques

STUDY DESIGN:
Intervention Model Description: We will include 152 medical students at the Universities of Bern, Fribourg and Zurich. Stratified by study site, students will be randomized to one of the two interventions. The blended-learning group will receive e-learning and near-peer tutoring over 16 weeks; the other group will receive 21 hours of teaching, from ultrasound experts, in a 2.5-day course.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blended learning (Experimental): Participants in the blended learning group will be taught abdominal ultrasound by an e-learning platform and practical near-peer tutoring classes over 16 weeks, summing up to 5 hours of e-learning and 16 hours of near-peer tutoring classes.
  Interventions: Other: Blended learning
- Standard course (Active Comparator): Participants in the standard course or control group will participate in a 2.5-day course in abdominal ultrasound, comprising 5 hours of lectures and 16 hours of ultrasound training.
  Interventions: Other: Standard course

INTERVENTIONS:
Other: Blended learning — In the intervention group, students will be given access to an e-learning platform that contains five e-learning modules. They will attend individual small group tutoring sessions, with a maximum of 4 students per group. They will be able to book these sessions at a dedicated web platform. They will have 16 weeks in which to complete the 5 e-learning modules and 16 hours of practical training. Progress will be monitored and supported by regular follow-up messages and calls by the study team. Students must hand in the logbook with tutors' signatures when they enter the exam. All students within the blended learning group that completed 5 hours of e-learning as well as 16 hours of peer-tutoring and passed a predefined total score in the test directly after the intervention will receive a course certificate. Students not fulfilling all of these criteria will have the possibility to complete the program and/or re-do the test after the end of the study.
  Arms: Blended learning
Other: Standard course — In the standard course or control group, students will participate in a 2.5-day course in abdominal ultrasound, comprising 5 hours of lectures and 16 hours of ultrasound training in small groups, with a maximum of 4 students per group. The course will be held in an ultrasound training centre in Bern. All students within the standard course group that participated in the whole 2.5 day course and passed a predefined total score in the test directly after the intervention will receive a course certificate. Students not fulfilling all of these criteria will have the possibility to complete the program and/or re-do the test after the end of the study.
  Arms: Standard course

SUMMARY:
Background:

Ultrasound has become clinical skill widely used in most medical disciplines. Institutions are changing their curricula to implementing basic ultrasound knowledge, often supplementing traditional teaching with 'near-peer' tutoring through classes held by advanced peers. Near-peer tutoring has been found to be both effective and cost-effective.

In Switzerland the most popular course in postgraduate training is a resource-intensive 21-hour basic course for abdominal ultrasound. However, this is expensive, and may not be the best way to impart these skills to undergraduates, who need training more adapted to their needs.

Therefore a 21-hour blended-learning ultrasound course, comprising 5 hours of e-learning and 16 hours of near-peer tutoring has been developped. Students and their near-peer tutors autonomously organize individual practical teaching sessions within a 16 weeks time period.

Methods:

Medical students from second to fourth year at the Universities of Bern, Fribourg and Zurich will be included. Stratified by study site, students will be randomized to one of the two interventions. The blended-learning group will receive e-learning and near-peer tutoring over 16 weeks; the other group will receive 21 hours of teaching, from ultrasound experts, in a 2.5-day course. All participants will undergo a six-station OSCE directly after the course and 6 months later. Students will fill out online questionnaires at baseline, directly after the course and 6 months later. The mean scores of both groups will be compared at six months after the end of both courses. Secondary outcome measures will be students' ultrasound skills immediately after the courses, student satisfaction, multivariate regression exploring factors that affect outcome at 6 months and exploratory subgroup analysis.

Discussion:

This study is designed to compare the current way of ultrasound education in Switzerland with a new blended learning course. It aims to determine whether the blended learning course is as good as, or better than the existing 21-hour standard course. If this is found to be the case, blended learning could help to expand capacity to offer such courses to undergraduate medical students. It would eventually allow undergraduate Swiss medical students to acquire ultrasound skills before starting their residencies. This study also aims at improving the understanding of how to achieve effective student-centred learning supported by near-peer tutoring.

DETAILED DESCRIPTION:
Background:

Over the last decades, ultrasound (US) examination has become commonly used in many medical specialties, including internal medicine and primary care. Young doctors often perform simple ultrasound investigations as residents in internal medicine or primary care especially in emergency care. Currently, 30% of Swiss primary care practices are equipped with an ultrasound machine.

The Swiss Society for Ultrasound in Medicine (SGUM/SSUM) is the accreditation body for ultrasound education in Switzerland. Doctors must obtain a certificate from the SGUM before they can bill ultrasound examinations for insurance payments. However, ultrasound courses are time-intensive (63 hours total, plus a final examination), and are offered in the postgraduate phase, when doctors often have few resources and little time. This may explain why only about half of General Practitioners who use ultrasound have the SGUM certificate. For the half without the certificate, not only can they not bill their ultrasound examination to an insurance company, but also the quality of the examination is less assured, as they have not demonstrated their competence in US skills in the SGUM examination. This may lead to insecurity for the patient and for the performing doctor. There is also a risk that this results in unnecessary examinations.

The SGUM certificate is achieved by passing three courses (basic/advanced/final; 21 hours each) as well as a summative final examination. Between courses, trainees must perform a certain number of US examinations on real patients, under direct and distant supervision. These courses are now being opened to undergraduates, and the 2017 revision of the Swiss learning objectives for medical studies (PROFILES) added basic US skills as mandatory learning goal.

In the past years US training courses at Swiss medical universities were mostly optional, and were quickly overbooked. This shortage of courses could be addressed by using near-peer tutors, which are increasingly used in faculty-organized US classes. Near-peer tutors are "trainees one or more years senior to trainees on the same level of medical education spectrum". Five randomized-controlled trials of ultrasound training have compared near-peer tutoring with faculty-led teaching and assessed students' practical ultrasound skills as a primary outcome measure. Four of these found peer-tutoring to be non-inferior and one found that students in the near-peer-tutoring group slightly underperformed.

Near-peer tutoring in undergraduate US training offers many potential advantages over traditional faculty-based teaching:

* Since mostly reciprocal US is being done by the participating medical students, perfect conditions for learning basic sonographic anatomy can be found. Medical students, in contrast to patients, are mostly slender, healthy and mobile.
* In near-peer tutoring settings, students are more likely to ask questions and participate actively. In addition, having ultrasound skills can help students feel more secure in their basic clinical examination skills.
* Near-peer tutoring relieves pressure on the university by alleviating the increasing teaching demand and by being cost-effective.
* There is evidence that students who work as tutors constantly improve their own skills.

In Autumn 2017, the Institute of Primary Health Care (BIHAM) at the University of Bern set up a working group of 24 US experts from all Swiss universities and of representatives of SGUM sections. The group decided on the "Swiss standard" for basic abdominal ultrasound examination after discussing it at two consensus-building meetings. In Spring 2018, videotapes of SGUM experts demonstrating the ultrasound examination of the various abdominal organs, based on that consensus, were recorded. These videos were integrated into interactive e-learning modules. They have been available to all Swiss medical students since the beginning of 2019.

In parallel, a formal system of training and continuous education for near-peer tutors was put in place by a collaboration of motivated students and faculty staff. Near-peer tutors receive at least 6 days of US training, including teaching on didactic techniques, and afterwards be registered as so-called 'junior-tutors' by SGUM. They must offer at least four hours of US class per semester, but can choose the times and dates. Tutors will be reimbursed for their teaching through course fees paid by course participants.

Methods:

The standard "Basic course in abdominal ultrasound", delivered over 2.5 consecutive days, contains 5 hours of theory and 16 hours of practical training. In contrast, our blended-learning course is more student-centred, in that it expects students to take the initiative to learn the theory from (A) the e-learning developed by the working group, and (B) 16 hours of near-peer tutoring in groups of two to four, at times that are mutually agreeable for tutors and students, without faculty involvement.

The e-learning is made up of five modules starting by an introductory e-learning module on technical basics in ultrasound, followed by four practical modules comprising the abdominal organs. For each of the four practical modules, students start by working through the e-learning module, followed by four hours of individual near-peer tutoring sessions.

Students decide the pace of their 16 hours of training, typically over a four-month period. When a student completes all five e-learning modules and has gathered 16 signatures from the peer-tutored classes, they can apply to take a summative final examination. If they pass the Objective Structured Clinical Examination (OSCE) validated by Hofer et al. (2011) and adapted to Swiss needs, they are accredited by SGUM, according to Swiss national accreditation guidelines, for the "Basic course in abdominal ultrasound" - the first of the three ultrasound courses within the SGUM curriculum.

The OSCE will be assessed twice for every participant. Once at the end of the course and once 6 months after the end of the course. The second OSCE will be the primary outcome, since it evaluates long-term retention of acquired US knowledge. Every student will be tested by six different examiners in each OSCE. Differences in difficulty of the four series of OSCE stations as well as difficulty of every station will be taken into account in the statistical analysis.

The blended-learning course offers several other advantages by implementing modern didactics: by distributing teaching sessions over 16 weeks instead of just 2.5 consecutive days, students benefit from "spaced repetition" which improves long term retention. In our programme, students can decide which session to choose next, and tutors and students arrange the teaching sessions according to their availability and needs, so learning is student-centred. These factors differentiate our study from the near-peer tutoring in ultrasound education reported in some studies, in which tutors engage in scheduled courses organized by university faculty.

Between randomization and the end of the training (t = 16 weeks), students will be instructed not to undergo any additional training (e-learning, practical sessions or other) other than those provided within the intervention. Additional training will be recorded directly after the end of the training by questionnaire and by going through e-learning logs. During the 6-month follow-up period, students in both groups will be equally encouraged to continue self-organised training and both will be granted access to ultrasound machines.

Adjusting to local curricula we will primarily recruit students in semester 7 in Bern (total medical student intake per year = 220) and in semester 6 in Zurich (240) and Fribourg (120). At each site, we will present the programme during a plenary session, assisted by our local co-investigators.

To avoid systematic differences in additional training during the follow-up period, the following rules will put in place:

* Students will only be told their test results from the first test after the end of the study
* Test performance in the follow-up test will have no effect on the accreditation

To reduce loss to follow-up, we will:

* Require all students who apply for the programme to sign a separate form confirming their availability and intention to complete the course and the examinations
* Reimburse participants 50.- CHF after they have taken the second OSCE.
* Reimburse travel costs for the second OSCE
* Hand out the test result and the course certificate only after the second OSCE

Students' motivation for ultrasound training is very high. The optional courses at Swiss universities are typically overbooked within minutes and many students are disappointed that they are unable to take part. Our study will give students the opportunity to get a certificate accredited by the SGUM for a course fee of 200.- CHF, regardless of the intervention they are assigned to. Postgraduate training for the same degree costs around 1200.- CHF.

We will use centralized computed randomization in blocks of 4 to allocate each of the participants to one of the two study arms, with allocation in a 1:1 ratio, stratified by study site. The reason for block randomisation is the requirement of the control group to comprise of exactly 24 or 28 students due to the maximum group size of 4 students per tutor. The randomization will be performed by a blinded external partner (Clinical Trials Unit in Bern).

Outcome assessors will be experienced sonographers who have not taught course participants of either group.

To ensure high interrater-reliability, faculty training for all assessors will be held immediately before the OSCE. In the first part of this training, the assessors discuss key aspects of the rating using videotaped examples of OSCE stations to achieve a common standard. At the end of the training, assessors will rate another video example, where the interrater-reliability will be assessed.

OSCE assessors will be blinded to group allocation. The assessments will be at the same time for each group. We will instruct students not to reveal their group allocation to the OSCE assessors.

Sample size calculation has been done as follows: Based on a pilot with 20 students we expect a mean score of 33/50 points per station with a standard deviation (SD) of 4 points. The study was powered for non-inferiority using a margin of a -1.5 points for the difference in mean OSCE scores between the intervention and control group in the practical exam at 6 months (primary outcome). 1.5 points difference would correspond to an effect size of 0.375 standard deviations (SD), which we would still consider as non-inferior. We calculated the sample size with the assumption that the intervention group will perform somewhat better (+0.5 in mean score) than the control group based on test results from previous pilots. We chose a 1-sided alpha-error of 0.05 and a power of 90% (138 participants). Allowing for a 9% dropout rate we decided to include 152 students.

Discussion:

If the new blended-learning format is shown to be at least as good as the existing standard course, we could quickly expand our capacity to offer such courses to undergraduate medical students, replacing resource-intensive faculty-led courses with peer-assisted learning programmes. This will eventually allow all undergraduate students to acquire ultrasound skills that will help them in their residencies. The national accreditation body fully supports this near-peer-tutoring-based course both financially and through full accreditation of a pilot project and has committed to continue its support if we find that this teaching format produces results that are just as good as, or better than, the usual faculty-led courses. Learning more about the advantages conferred by student-centred learning through near-peer teaching will enable us to design better peer-assisted learning programmes and to design new, similar programmes in other areas.

ELIGIBILITY:
Inclusion Criteria:

* Medical students at three Swiss universities (Bern, Freiburg, Zurich) in the 3rd to 8th semester, who:
* are willing to participate in the study;
* are willing to pay the 200.- CHF course fees (partial reimbursement of tutors and administrative fee for the SGUM course certificate)
* fill out a baseline questionnaire
* signed informed consent sheet

Exclusion Criteria:

* Did not sign study agreement or pay the course fee
* More than 5 hours of previous formal ultrasound training
* Failure to fill out baseline questionnaire

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2021-11-21 (Actual)

PRIMARY OUTCOMES:
Mean participants' "Swiss Students' Ultrasound Skills Assessment" scores six months after the end of their courses (OSCE 2). | 10 months from enrollment at each site
  The investigators will assess the participants' ultrasound skills using the "Swiss Students' Ultrasound Skills Assessment". This uses a validated OSCE form (Hofer et al. 2011), which has been adapted to specific Swiss needs and revalidated. The total score can range from 0-300 points, a higher total representing a better performance. The OSCE assesses handling of the probe, explanation of the ultrasound image, examination skills and theoretical knowledge. Each station will assess a key topic that arises in both courses.

SECONDARY OUTCOMES:
Mean participants' "Swiss Students' Ultrasound Skills Assessment" scores immediately after the end of their courses (OSCE 1). | 16 weeks from enrollment at each site
  As above.
Change in mean participants' "Swiss Students' Ultrasound Skills Assessment" scores (knowledge retention). | 10 months from enrollment at each site
  To evaluate knowledge retention, the investigators will analyse the change in mean "Swiss Students' Ultrasound Skills Assessment" scores between the end of the courses and 6 months later,
Participants' satisfaction with allocated courses | 16 weeks from enrollment at each site
  Students will complete a "Ultrasound Course Satisfaction Rating Scale" questionnaire immediately before OSCE 1. This will assess participants' satisfaction with their respective courses, through their mean Likert scale scores (Possible scores for each question 1-5, where 1 = Very dissatisfied, 5 = Very satisfied).
Multivariate regression exploring factors that affect outcome at six months after the end of their courses | 10 months after enrollment at each site
  The investigators will use multivariate regression to explore factors that affect the outcome at 6 months after the end of the courses (e.g. group allocation, additional hours of self-training, average group size during training, gender).

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hari, MD, Principal Investigator — University of Bern
Locations (3):
- Switzerland (3):
  - University of Bern, Bern
  - University of Fribourg, Fribourg
  - University of Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bornemann P, Barreto T. Point-of-Care Ultrasonography in Family Medicine. Am Fam Physician. 2018 Aug 15;98(4):200-202. No abstract available. PMID 30215979
- [Background] Ultrasound Guidelines: Emergency, Point-of-Care and Clinical Ultrasound Guidelines in Medicine. Ann Emerg Med. 2017 May;69(5):e27-e54. doi: 10.1016/j.annemergmed.2016.08.457. No abstract available. PMID 28442101
- [Background] Ma IWY, Arishenkoff S, Wiseman J, Desy J, Ailon J, Martin L, Otremba M, Halman S, Willemot P, Blouw M; Canadian Internal Medicine Ultrasound (CIMUS) Group*. Internal Medicine Point-of-Care Ultrasound Curriculum: Consensus Recommendations from the Canadian Internal Medicine Ultrasound (CIMUS) Group. J Gen Intern Med. 2017 Sep;32(9):1052-1057. doi: 10.1007/s11606-017-4071-5. Epub 2017 May 11. PMID 28497416
- [Background] Rikley E, Boillat-Blanco N, Meuwly JY, Breuss E, Senn N. [Ultrasonography : an useful diagnostic tool for the general practitioner]. Rev Med Suisse. 2017 Mai 10;13(562):990-994. French. PMID 28627842
- [Background] Hoppmann RA, Rao VV, Bell F, Poston MB, Howe DB, Riffle S, Harris S, Riley R, McMahon C, Wilson LB, Blanck E, Richeson NA, Thomas LK, Hartman C, Neuffer FH, Keisler BD, Sims KM, Garber MD, Shuler CO, Blaivas M, Chillag SA, Wagner M, Barron K, Davis D, Wells JR, Kenney DJ, Hall JW, Bornemann PH, Schrift D, Hunt PS, Owens WB, Smith RS, Jackson AG, Hagon K, Wilson SP, Fowler SD, Catroppo JF, Rizvi AA, Powell CK, Cook T, Brown E, Navarro FA, Thornhill J, Burgis J, Jennings WR, McCallum JB, Nottingham JM, Kreiner J, Haddad R, Augustine JR, Pedigo NW, Catalana PV. The evolution of an integrated ultrasound curriculum (iUSC) for medical students: 9-year experience. Crit Ultrasound J. 2015 Dec;7(1):18. doi: 10.1186/s13089-015-0035-3. Epub 2015 Nov 21. PMID 26589313
- [Background] Education and Practical Standards Committee, European Federation of Societies for Ultrasound in Medicine and Biology. Minimum training recommendations for the practice of medical ultrasound. Ultraschall Med. 2006 Feb;27(1):79-105. doi: 10.1055/s-2006-933605. No abstract available. PMID 16508866
- [Background] Wakefield RJ, Weerasinghe A, Tung P, Smith L, Pickering J, Msimanga T, Arora M, Flood K, Gupta P, Bickerdike S, McLaughlan J, Uttley A, Wilson J, Evans T, Wolstenhulme S, Roberts TE. The development of a pragmatic, clinically driven ultrasound curriculum in a UK medical school. Med Teach. 2018 Jun;40(6):600-606. doi: 10.1080/0142159X.2018.1439579. Epub 2018 Feb 28. PMID 29490531
- [Background] Bulte C, Betts A, Garner K, Durning S. Student teaching: views of student near-peer teachers and learners. Med Teach. 2007 Sep;29(6):583-90. doi: 10.1080/01421590701583824. PMID 17922356
- [Background] Celebi N, Zwirner K, Lischner U, Bauder M, Ditthard K, Schurger S, Riessen R, Engel C, Balletshofer B, Weyrich P. Student tutors are able to teach basic sonographic anatomy effectively - a prospective randomized controlled trial. Ultraschall Med. 2012 Apr;33(2):141-5. doi: 10.1055/s-0029-1245837. Epub 2010 Nov 23. PMID 21104601
- [Background] Knobe M, Munker R, Sellei RM, Holschen M, Mooij SC, Schmidt-Rohlfing B, Niethard FU, Pape HC. Peer teaching: a randomised controlled trial using student-teachers to teach musculoskeletal ultrasound. Med Educ. 2010 Feb;44(2):148-55. doi: 10.1111/j.1365-2923.2009.03557.x. Epub 2009 Dec 21. PMID 20040056
- [Background] Knobe M, Sellei RM, Maus U, Mooij SC, Gradl G, Sopka S, Niethard FU, Pape HC. [Undergraduate curricular training in musculoskeletal ultrasound: the impact of preexisting anatomic knowledge]. Z Orthop Unfall. 2010 Dec;148(6):685-90. doi: 10.1055/s-0030-1250378. Epub 2010 Oct 12. German. PMID 20941690
- [Background] Kuhl M, Wagner R, Bauder M, Fenik Y, Riessen R, Lammerding-Koppel M, Gawaz M, Fateh-Moghadam S, Weyrich P, Celebi N. Student tutors for hands-on training in focused emergency echocardiography--a randomized controlled trial. BMC Med Educ. 2012 Oct 29;12:101. doi: 10.1186/1472-6920-12-101. PMID 23107588
- [Background] Garcia-Casasola G, Sanchez FJ, Luordo D, Zapata DF, Frias MC, Garrido VV, Martinez JV, de la Sotilla AF, Rojo JM, Macho JT. Basic Abdominal Point-of-Care Ultrasound Training in the Undergraduate: Students as Mentors. J Ultrasound Med. 2016 Nov;35(11):2483-2489. doi: 10.7863/ultra.15.11068. Epub 2016 Oct 13. PMID 27738292
- [Background] Ten Cate O, Durning S. Peer teaching in medical education: twelve reasons to move from theory to practice. Med Teach. 2007 Sep;29(6):591-9. doi: 10.1080/01421590701606799. PMID 17922354
- [Background] Garcia de Casasola Sanchez G, Gonzalez Peinado D, Sanchez Gollarte A, Munoz Aceituno E, Pena Vazquez I, Torres Macho J. Teaching of clinical ultrasonography to undergraduates: students as mentors. Rev Clin Esp (Barc). 2015 May;215(4):211-6. doi: 10.1016/j.rce.2014.11.023. Epub 2015 Jan 10. English, Spanish. PMID 25583252
- [Background] Dietrich CF, Hoffmann B, Abramowicz J, Badea R, Braden B, Cantisani V, Chammas MC, Cui XW, Dong Y, Gilja OH, Hari R, Nisenbaum H, Nicholls D, Nolsoe CP, Nurnberg D, Prosch H, Radzina M, Recker F, Sachs A, Saftoiu A, Serra A, Sweet L, Vinayak S, Westerway S, Chou YH, Blaivas M. Medical Student Ultrasound Education: A WFUMB Position Paper, Part I. Ultrasound Med Biol. 2019 Feb;45(2):271-281. doi: 10.1016/j.ultrasmedbio.2018.09.017. Epub 2018 Nov 27. PMID 30497768
- [Background] Raschle N, Hari R. [Blended Learning Basic Course Sonography - A SGUM Accredited Ultrasound Course Based on Peer-Tutoring]. Praxis (Bern 1994). 2018 Nov;107(23):1255-1259. doi: 10.1024/1661-8157/a003116. German. PMID 30424697
- [Background] Augustin M. How to learn effectively in medical school: test yourself, learn actively, and repeat in intervals. Yale J Biol Med. 2014 Jun 6;87(2):207-12. eCollection 2014 Jun. PMID 24910566
- [Background] Suresh K. An overview of randomization techniques: An unbiased assessment of outcome in clinical research. J Hum Reprod Sci. 2011 Jan;4(1):8-11. doi: 10.4103/0974-1208.82352. PMID 21772732
- [Background] Hofer M, Kamper L, Sadlo M, Sievers K, Heussen N. Evaluation of an OSCE assessment tool for abdominal ultrasound courses. Ultraschall Med. 2011 Apr;32(2):184-90. doi: 10.1055/s-0029-1246049. Epub 2011 Feb 14. PMID 21321843
- [Background] Lipsey MW, Wilson DB. The efficacy of psychological, educational, and behavioral treatment. Confirmation from meta-analysis. Am Psychol. 1993 Dec;48(12):1181-209. doi: 10.1037//0003-066x.48.12.1181. PMID 8297057
- [Background] Michaud PA, Jucker-Kupper P, The Profiles Working Group. The "Profiles" document: a modern revision of the objectives of undergraduate medical studies in Switzerland. Swiss Med Wkly. 2016 Feb 1;146:w14270. doi: 10.4414/smw.2016.14270. eCollection 2016. PMID 26829005